CLINICAL TRIAL: NCT06789159
Title: A Phase Ib Study of VK-2019 in Patients With Relapsed or Refractory EBV+ Diffuse Large B-cell Lymphomas (DLBCL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Wistar Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2024-0941; R01CA282411 (NIH); JT 35884 (Other: JeffTrial Number)
Record Dates: First submitted 2025-01-02; First posted 2025-01-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B Cell Lymphoma Refractory; Diffuse Large B Cell Lymphoma Relapsed; Epstein-Barr Virus (EBV) Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment (VK-2019 Dose 600mg) (Experimental): Dose cohort A will dose at 600mg. VK-2019 will be administered daily starting on day 1 of cycle 1 (D1C1). Dose cohort A will dose at 600 mg dose. Treatment cycles will repeat every 28 days , in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: VK-2019
- Treatment (VK-2019 Dose 1200mg) (Experimental): Dose cohort B will dose at 1200mg.VK-2019 will be administered daily starting on day 1 of cycle 1 (D1C1). Dose cohort B will dose at 1200 mg dose. Treatment cycles will repeat every 28 days , in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: VK-2019
- Treatment (VK-2019 Dose 1800mg) (Experimental): Dose cohort C will dose at 1800mg. VK-2019 will be administered daily starting on day 1 of cycle 1 (D1C1). Dose cohort C will dose at 1800 mg dose. Treatment cycles will repeat every 28 days , in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: VK-2019

INTERVENTIONS:
Drug: VK-2019 — VK-2019 will be administered daily starting on day 1 of cycle 1 (D1C1). Dose cohort A will dose at 600 mg dose cohort B 1200 mg and dose cohort C 1800 mg. Treatment cycles will repeat every 28 days , in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This is a Phase Ib in adult patients with relapsed or refractory EBV-positive DLBCL using daily oral dosing of VK-2019 in three dose escalation cohorts: 600 mg/day, 1200 mg/day, 1800 mg/day for 28 days (cycle), until progression or toxicity.

DETAILED DESCRIPTION:
This is an open label, dose-escalation phase Ib study with biomarker assessments to determine the safety and tolerability of single agent VK-2019 in patients with relapsed or refractory EBV-positive lymphomas.

Each treatment cycle is comprised of a daily dose of VK-2019 administered orally for 28 days with a response assessment every 3 cycles. All subjects will be monitored for survival for 3 years.

VK-2019 will be administered daily starting on day 1 of cycle 1 (D1C1). Dose cohort A will dose at 600 mg dose cohort B 1200 mg and dose cohort C 1800 mg. Treatment cycles will repeat every 28 days , in the absence of disease progression or unacceptable toxicity. Should dose cohort 1 result in unacceptable toxicity, the protocol will be amended to include a dose (-1) cohort of VK-2019 given in the same fashion as above.

Patients who achieve at least stable disease (SD, PR, or CR) after completing 3 cycles can continue receiving therapy. Patients who have progressive disease (PD) after cycle 3 will discontinue protocol treatment. All patients will be followed for a total of 3 years.

Protocol therapy will be discontinued at any time if a patient withdraws consent, has progressive disease, unacceptable toxicity, or pregnancy is suspected.

ELIGIBILITY:
4.1 Inclusion Criteria

1. Informed consent obtained prior to any protocol mandated assessment.
2. Age ≥ 18 years.
3. Patient must have relapsed or refractory EBV-positive DLBCL after a minimum of 2 prior regimens of systemic therapy.
4. Patient must have exhausted all available standard of care treatment options that could potentially provide clinical benefit.
5. Toxicities related to prior therapy must have returned to Grade 1 or less, or if chronic must be stable. Peripheral neuropathy must be Grade 2 or less
6. Prior anti-cancer treatment must have been completed greater than 2 weeks prior to study day 1.
7. Patients must have measurable disease, as defined by IWG 2007 criteria.
8. ECOG performance status score of ≤2
9. Adequate organ function as defined by the following criteria:

   1. Absolute neutrophil count > 1,500/microl (stable off any growth factor within 1 week of study drug administration)
   2. Hemoglobin > 9 g/dL (transfusion to achieve this level is permitted)
   3. Platelet count > 75,000/microl (transfusion to achieve this level is NOT permitted)
   4. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN);
   5. Total serum bilirubin ≤ 1.5 x ULN;
   6. Creatinine clearance≥ 60 ml/min as calculated per Cockcroft and Gault equation.
   7. Urinary protein < 2+ by dipstick. If dipstick ≥ 2+, then a 24-hour urine collection can be done, and the patient may enter only if urinary protein is < 1 g/24 hour;
10. Sexually active patients will agree to utilize birth control method during the study and for 18 weeks after the study is concluded, using effective birth control methods as defined in https://www.cdc.gov/reproductivehealth/unintendedpregnancy/pdf/contraceptive_methods_508.pdf. See Protocol Appendix C.
11. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

4.2 Exclusion Criteria

1. Patients with severe or active symptomatic cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease within the last 12 months; chronic obstructive pulmonary disease exacerbation other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders; patents with effectively treated conditions (e.g. stenting for CAD) are eligible.
2. Patients with metastatic disease with active central nervous system (CNS) involvement, defined as parenchymal brain or leptomeningeal involvement.
3. Concurrent administration of herbal preparations.
4. A serious uncontrolled medical disorder or active infection which would impair the ability of the subject to receive protocol therapy or whose control may be jeopardized by the complications of this therapy.
5. Patients currently taking drugs that inhibit or induce OATP1B1 or OATP1B3 within 5 half- lives of that agent. Examples are included in Appendix B.
6. Patients currently taking drugs that are proton pump inhibitors (PPIs) within 5 half- lives of that agent. Examples are included in Appendix B.
7. Patients who have received a prior organ allograft or allogeneic bone marrow transplant are eligible but must have no evidence of active GVHD and be off immunosuppressive drugs.
8. Current non-prescription drug or alcohol dependence;
9. For all female patients, pregnancy or breastfeeding.
10. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.
12. Patients with corrected QT by Fridericia's formula (QTcF) of >470 ms are excluded.
13. Patients with Post-Transplant Lymphoproliferative Disease (PTLD) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety Dose- Maximum Tolerated Dose | At the end of Cycle 1 (each cycle is 28 days), until disease progression or unacceptable toxicity. All Patients will be followed for a total of 3 years.
  • The maximum tolerated dose (MTD) of single agent VK-2019 based upon treatment emergent AE (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wysota, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (1):
- Honickman Center, Philadelphia, Pennsylvania, United States